CLINICAL TRIAL: NCT03459144
Title: Comparison of the Effects of Photodynamic Therapy, Intravitreal Ranibizumab and Combination for Polypoidal Choroidal Vasculopathy Under 1+PRN Regimen
Brief Title: Comparison of PDT, Intravitreal Ranibizumab and Combination for Polypoidal Choroidal Vasculopathy Under 1+PRN Regimen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Chen-jin, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017KYPJ093
Record Dates: First submitted 2018-02-27; First posted 2018-03-08 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Polypoidal Choroidal Vasculopathy
Keywords: polypoidal choroidal vasculopathy; photodynamic therapy; ranibizumab; combination therapy; cost-benefit
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy | interventions — Verteporfin; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- photodynamic therapy (Experimental): Participants will be given the standard verteporfin photodynamic therapy at baseline followed by additional standard verteporfin PDT as needed (every three months)(namely 1+PRN regimen).
  Interventions: Drug: verteporfin; Drug: verteporfin and ranibizumab
- intravitreal ranibizumab (Experimental): Participants will receive the intravitreal ranibizumab treatment (0.05mg) at baseline and additional intravitreal ranibizumab will be given to the participants when necessary (every month) (namely 1+PRN regimen).
  Interventions: Drug: verteporfin; Drug: verteporfin and ranibizumab
- combination therapy of PDT and IVR (Experimental): Participants will be given the standard verteporfin photodynamic therapy followed by intravitreal ranibizumab (0.05mg) 72h after the standard verteporfin PDT treatment at baseline. Additional verteporfin photodynamic therapy and intravitreal ranibizumab (0.05mg) will be given to the participants when necessary (every month)(namely 1+PRN regimen).
  Interventions: Drug: verteporfin; Drug: verteporfin and ranibizumab

INTERVENTIONS:
Drug: verteporfin — Participants will receive the intravitreal ranibizumab treatment (0.05mg) at baseline and additional intravitreal ranibizumab(0.05mg) will be given to the participants when necessary（every three months）.
  Other Names: ranibizumab
Drug: verteporfin and ranibizumab — Participants will be given the standard verteporfin photodynamic therapy followed by intravitreal ranibizumab (0.05mg) 72h after the PDT treatment at baseline. Additional verteporfin photodynamic therapy and intravitreal ranibizumab (0.05mg) will be given to the participants when necessary.

SUMMARY:
The aim of this study is to compare the outcomes of different treatment methods including photodynamic therapy (PDT), intravitreal ranibizumab injection (IVR) and combination therapy under the "1+PRN" treatment regimen for polypoidal choroidal vasculopathy (PCV) and find the optimal treatment for PCV.

DETAILED DESCRIPTION:
The optimal treatment for PCV is still under debate. Little knowledge is known about the treatment effect of "1+pro re nata(PRN)" treatment regimen for PCV. The aim of this study is to compare the outcomes of different treatment methods including PDT, IVR and combination therapy under the "1+PRN" treatment regimen for PCV.

The study is the first prospective randomized controlled trial about different treatment methods on PCV under "1+PRN" treatment regimen. The null hypothesis of the study is that combination therapy may be the optimal treatment method for PCV. The primary outcome measures is the Best-corrected visual acuity (BCVA) of the participants at 1 year after treatment. Besides, the slit-lamp examination, tonometry, funduscopy, and OCT, FFA, ICGA examinations will also be compared between different groups to find the optimal treatment for PCV.

ELIGIBILITY:
Inclusion Criteria:

1. active macula-involved polypoidal lesions evidenced by ICGA;
2. greatest linear dimension of 5400 μm or less assessed by ICGA;
3. follow-up of at least 12 months.

Exclusion Criteria:

1. any other ocular disease, such as ocular trauma, glaucoma, uveitis, diabetic retinopathy, angioid streaks, pathologic myopia, or presumed ocular histoplasmosis syndrome;
2. any systemic contraindication to the PDT, IVR, sodium fluorescein, or indocyanine green dyes;
3. any severe uncontrolled systemic disease, such as uncontrolled hypertention, coronary heart disease, liver failure, or kidney failure.

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2015-07-30 (Actual); Study Completion 2015-07-30 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity | 12 months
  the best corrected visual acuity is the Primary Outcome Measure

CONTACTS AND LOCATIONS:
Overall Officials: Chenjin Jin, Ph.D., Study Chair — State Key Laboratory of Ophthalmology, Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lai K, Li Y, Zhou L, Zhong X, Huang C, Xu F, Lu L, Ge J, Jin C. Comparison of the effects of photodynamic therapy, intravitreal ranibizumab and combination for polypoidal choroidal vasculopathy under 1 + PRN regimen. BMC Ophthalmol. 2018 Jun 20;18(1):144. doi: 10.1186/s12886-018-0801-7. PMID 29925341